CLINICAL TRIAL: NCT04293016
Title: Building Resilience In Caregivers of Trauma Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah M Little, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-19-0073
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Caregiver Burnout
Keywords: PTSD; Depression; substance use
MeSH Terms: conditions — Caregiver Burden; Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Support as usual (Active Comparator)
  Interventions: Behavioral: Support as usual
- Problem Solving therapy (Experimental)
  Interventions: Behavioral: Problem solving therapy
- ICU diary (Experimental)
  Interventions: Behavioral: ICU diary

INTERVENTIONS:
Behavioral: Support as usual — This group receives current best practice which includes participation in ICU support groups and provision of community support resources
  Arms: Support as usual
Behavioral: Problem solving therapy — This group will receive one on one therapy based on identifying stressors and solutions to those stressors
  Arms: Problem Solving therapy
Behavioral: ICU diary — This group will be provided with a structured written diary that includes identification of stressors and development of solutions to those stressors
  Arms: ICU diary

SUMMARY:
The purpose of the study is to examine the role of demographics, pre-existing anxiety, depression, and substance use on caregiver depression anxiety, and substance use following a critical injury to a loved one, evaluate the factors that mediate the effectiveness of traditional psychotherapy using problem solving therapy to reduce depression, anxiety, and substance use and to evaluate the factors that mediate the effectiveness of providing an ICU diary and instruction on that diary to reduce depression, anxiety, and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Must anticipate serving in a Caregiver role after the patient is discharged (A. Must be either a family member or close friend of a patient who has been admitted to the trauma/critical care service ICU B. Must anticipate spending time with the patient in a caregiver or other supportive role (e.g., emotional, social, financial) after the patient is discharged
* Caregiver and patient must report English as a primary language
* Patient and Caregiver must be able to provide informed consent
* Caregiver must be able to provide at least two forms of contact information
* Trauma Patient directly admitted to the ICU (Primary cause of admission is trauma, Injury must include trauma to the head/brain or polytrauma, Admitted directly to the hospital, Patient admission of at least 48 hours, Patient is currently admitted to the ICU, Patient is expected to survive more than 96 hours at 48 hours after admission, Patient has an abbreviated injury score greater than 3 (severe, critical, maximum), Fluent in English)
* Trauma patient must be able to communicate verbally

Exclusion

* Does not anticipate serving in a Caregiver role after the patient is discharged
* Caregiver is not a close friend or family member of the patient who has been admitted to the ICU
* Caregiver does not expect to serve in a supportive role to the patient
* Caregiver does not meet inclusion criteria as stated above
* Patient is not currently admitted to the ICU and or is not expected to remain in the ICU for 48 hours
* Patient is not expected to survive more than 96 hours
* Patient is not expected to require assistance prior to discharge
* Patient is not between 17 and 65 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-18 (Estimated); Study Completion 2024-08-26 (Estimated)

PRIMARY OUTCOMES:
Short form survey (SF-12) | 6 months post injury
  Quality of life of caregiver as assessed by the short form survey (SF-12).The SF-12 is a 12 item questionnaire with a range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Posttraumatic Stress Disorder Checklist (PCL-5) | 6 months post injury
  The extent to which caregivers have been bothered by PTSD symptoms as assessed by the PTSD Checklist (PCL-5) assessment.The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The Hamilton Depression Rating Scale (HAM-D) | 6 months post injury
  Symptoms of depression in caregivers as assessed by the The Hamilton Depression Rating Scale (HAM-D).Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0(Absent)-2(frequent)

SECONDARY OUTCOMES:
The center for epidemiologic studies of depression (CESD-R ) | 3 months post injury
  Depression in caregivers as assessed by the CESD-R tool The CESD-R scale has 20 items and each is measured from 0(not at all) to 4(nearly every day for 2 weeks)
PTSD Checklist for (PCL-5) assessment. | 3 months post injury
  The extent to which caregivers have been bothered by PTSD symptoms as assessed by the PTSD Checklist (PCL-5) assessment.The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past month (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely).
The Alcohol Use Disorders identification Test (AUDIT): | 3 months post injury
  Alcohol use problems in caregivers as assessed by the AUDIT scale This is a 10-item screening tool and is rated between 0-4-the higher number indicating a worse outcome
Number of days of hospitalization | 6 months post injury
  Medical record based review of hospital readmission
Number of infections post discharge | 6 months post injury
  Medical record based review of number of infections after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Little, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No